CLINICAL TRIAL: NCT02517294
Title: "Mucosal Injury During Nasotracheal Intubation for Dental Procedures in Children-does the Tube Design Matter?"
Brief Title: , "Mucosal Injury During Nasotracheal Intubation for Dental Procedures in Children-does the Tube Design Matter?"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: #15-17
Record Dates: First submitted 2015-05-22; First posted 2015-08-07 (Estimated); Results first posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Epistaxis
Keywords: Nasotracheal intubation; adenoid size; epistaxis; nasopharyngeal mucosal injury
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard nasotracheal tube (Active Comparator): Nasotracheal intubation using 'standard' side-beveled nasotracheal tubes
  Interventions: Device: Standard nasotracheal tube
- Parker flex-tip nasotracheal tube (Active Comparator): Nasotracheal intubation using 'experimental' flex-tip midline-beveled nasotracheal tubes
  Interventions: Device: Parker flex-tip nasotracheal tube

INTERVENTIONS:
Device: Parker flex-tip nasotracheal tube — specially designed nasotracheal tube used for nasotracheal intubation assess nasopharynx for severity of bleeding grade adenoid size
  Arms: Parker flex-tip nasotracheal tube
Device: Standard nasotracheal tube — standard nasotracheal tube for nasotracheal intubation assess nasopharynx for severity of bleeding grade adenoid size
  Arms: standard nasotracheal tube

SUMMARY:
Comparison is made between standard nasotracheal tubes and a specially designed nasotracheal tube during nasotracheal intubation in children undergoing general anesthesia for dental surgery.

DETAILED DESCRIPTION:
The Parker flex-tip, midline-beveled nasotracheal tube theoretically slides past obstruction in the nasopharynx causing less mucosal damage than standard nasotracheal tubes.

The investigators aim to test whether mucosal injury during nasotracheal intubation in children undergoing general anesthesia for dental procedures can thus be minimized taking into consideration adenoid size, and differences in nasopharyngeal diameter.

ELIGIBILITY:
Inclusion Criteria:

* children between the ages of 3-11, ASA 1-3, presenting to Wolfson Children's Hospital (WCH) for dental procedures requiring general anesthesia with nasotracheal intubation.

Exclusion Criteria:

* ASA >3
* known bleeding disorders
* recent or ongoing treatment with blood-thinning medicines
* frequent epistaxis
* active URI/congestion/rhinorrhea
* craniofacial abnormalities prohibiting NTI
* known difficult airway
* prior nasal surgery/trauma
* allergies to any of the medicines used in this study.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Bryskin, MD, Principal Investigator — Nemours Children's Clinic, Jacksonville, FL
Locations (1):
- Wolfson Children's Hospital, Jacksonville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Nasotracheal Tube | Parker Flex-tip Nasotracheal Tube
Started | 38 | 35
Completed | 38 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Nasotracheal Tube | Parker Flex-tip Nasotracheal Tube | Total
Number analyzed (Participants) | 38 | 35 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 38 | 35 | 73
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.13 (1.98) | 6.43 (2.20) | 6.27 (2.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 26 | 24 | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 38 | 35 | 73
BMI [Mean (Standard Deviation); unit: kg/m^2] | 16.9 (3.33) | 16.9 (4.46) | 16.9 (3.88)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Epistaxis
Description: Mucosal damage as quantified by presence and severity of bleeding immediately after passage of the NTT through the nasopharynx.
Time Frame: within approximately 4hrs of surgery (day of surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Nasotracheal Tube | Parker Flex-tip Nasotracheal Tube
Number analyzed (Participants) | 38 | 35
Participants | 11 | 2

2. Secondary Outcome: Number of Participants With Nasotracheal Tube Impingement
Description: Presence and degree of severe impingement of the nasotracheal tube during nasotracheal intubation
Time Frame: perioperative, immediate during intervention - expected 2hrs (day of surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Nasotracheal Tube | Parker Flex-tip Nasotracheal Tube
Number analyzed (Participants) | 38 | 35
Participants | 6 | 3

3. Secondary Outcome: Number of Participants With Postoperative Epistaxis
Description: ongoing nasal bleeding in the recovery unit
Time Frame: Participants will be followed for the duration of the hospital stay, an expected average of 6 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Nasotracheal Tube | Parker Flex-tip Nasotracheal Tube
Number analyzed (Participants) | 38 | 35
Participants | 1 | 0

4. Secondary Outcome: Number of Participants With Postoperative Croup
Description: evidence of glottic edema/injury in the immediate postoperative time frame
Time Frame: end of surgery until time of discharge, approximately 4hrs
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Nasotracheal Tube | Parker Flex-tip Nasotracheal Tube
Number analyzed (Participants) | 38 | 35
Participants | 0 | 1

5. Secondary Outcome: Time to Discharge in Minutes
Time Frame: emergence from anesthesia to meeting discharge criteria, approximately 4hrs
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Standard Nasotracheal Tube | Parker Flex-tip Nasotracheal Tube
Number analyzed (Participants) | 38 | 35
minutes | 32.1 (13.5) | 30.4 (10.8)

ADVERSE EVENTS:
Time Frame: day of procedure, up to 12 hours
Description: the study did not include experimental equipment or a deviation from the standard of care
Arm/Group | Standard Nasotracheal Tube | Parker Flex-tip Nasotracheal Tube
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/35
Other Adverse Events (participants affected / at risk) | 0/38 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-10): https://cdn.clinicaltrials.gov/large-docs/94/NCT02517294/Prot_SAP_000.pdf